CLINICAL TRIAL: NCT00002594
Title: Dose-Intensive Melphalan and Cyclophosphamide With Autologous Bone Marrow Rescue for Recurrent Medulloblastoma and Germ Cell Tumors
Brief Title: Combination Chemotherapy Followed by Bone Marrow and/or Peripheral Stem Cell Transplantation in Treating Patients With Recurrent Medulloblastoma or CNS Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9430; COG-P9430 (Other: Children's Oncology Group); POG-9430 (Other: Pediatric Oncology Group); CDR0000063784 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: recurrent childhood brain tumor; childhood central nervous system germ cell tumor; recurrent childhood medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Medulloblastoma | interventions — sargramostim; Macrophage Colony-Stimulating Factor; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Cyclophosphamide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablative chemo followed by autologous bone marrow (ABM) rescue (Experimental): Autologous bone marrow and/or peripheral blood stem cells (PBSC) are harvested. Patients then receive intensive cyclophosphamide IV over 1 hour on days -8 to -5 and melphalan IV over 15 minutes on days -4 to -2. Bone marrow is reinfused on day 0. PBSC are reinfused on day 0 if used alone or on day 1 if used after autologous bone marrow transplantation (ABMT). Sargramostim (GM-CSF) is administered IV over 2 hours daily beginning 4 hours after ABMT and continuing until blood counts recover.
  Interventions: Biological: Sargramostim; Drug: cyclophosphamide; Drug: melphalan; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: Sargramostim — Given IV
  Other Names: M-CSF; GM-CSF; Granulocyte macrophage-colony stimulating factor; Prokine; Leukine; NSC #6137
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC #026271; IND #7089
Drug: melphalan — Given IV
  Other Names: ylalanine mustard; L-PAM; L-sarcolysin; Alkeran; NSC #8806
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so that they stop growing or die. bone marrow transplantation and peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by bone marrow transplantation and/or peripheral stem cell transplantation in treating patients who have recurrent medulloblastoma or CNS germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response and progression-free survival in patients with recurrent medulloblastoma or CNS germ cell tumors treated with intensive melphalan and cyclophosphamide followed by autologous bone marrow and/or peripheral blood stem cell rescue.
* Determine the acute and delayed toxic effects of this regimen in these patients.

OUTLINE: Autologous bone marrow and/or peripheral blood stem cells (PBSC) are harvested. Patients then receive intensive cyclophosphamide IV over 1 hour on days -8 to -5 and melphalan IV over 15 minutes on days -4 to -2. Bone marrow is reinfused on day 0. PBSC are reinfused on day 0 if used alone or on day 1 if used after autologous bone marrow transplantation (ABMT). Sargramostim (GM-CSF) is administered IV over 2 hours daily beginning 4 hours after ABMT and continuing until blood counts recover.

Patients are followed every 6 months through year 4 and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent medulloblastoma or CNS germ cell tumor

  * Histologic review of the primary intracranial or spinal cord tumor required

    * Biopsy and reduction of tumor bulk prior to study encouraged but not required
* No more than 1 prior primary therapy (radiotherapy or chemoradiotherapy) and/or 1 prior salvage therapy

  * Patients with progression on salvage therapy ineligible
* Minimal residual disease (tumor bulk no more than 1.5 cm) or in second clinical complete remission (CR)
* Bone marrow infiltration with or without mass lesions or isolated abnormal CSF cytology as the only manifestation of recurrent disease allowed if a clinical CR is first achieved with conventional therapy

PATIENT CHARACTERISTICS:

Age:

* 2 to 25

Performance status:

* Karnofsky 80-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGPT less than 80 IU

Renal:

* Creatinine less than 1.2 mg/dL

Cardiovascular:

* LVEF normal

Other:

* No infection
* Able to tolerate vigorous hydration
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior cyclophosphamide or ifosfamide allowed

Endocrine therapy:

* No concurrent dexamethasone as an antiemetic
* Other concurrent corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* Pretransplantation radiotherapy boost allowed

Surgery:

* See Disease Characteristics
* Pretransplantation surgery allowed

Other:

* At least 4 weeks since prior therapy except corticosteroids

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 1994-09; Primary Completion 2003-09 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald H. Mahoney, MD, Study Chair — Texas Children's Cancer Center
Locations (118):
- United States (103):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Stanford University Medical Center, Stanford, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - Beth Israel Hospital North, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission St. Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Warren Clinic, Tulsa, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - East Tennessee State University Cancer Center at JCMC, Johnson City, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Result] Kadota RP, Mahoney DH, Doyle J, Duerst R, Friedman H, Holmes E, Kun L, Zhou T, Pollack IF. Dose intensive melphalan and cyclophosphamide with autologous hematopoietic stem cells for recurrent medulloblastoma or germinoma. Pediatr Blood Cancer. 2008 Nov;51(5):675-8. doi: 10.1002/pbc.21655. PMID 18623206